CLINICAL TRIAL: NCT01657968
Title: Procalcitonin-guided Detection of Streptococcal Acute Tonsillitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Skodstrup Medical Clinic, Denmark (Unknown)
Responsible Party: Principal Investigator, Ann Christensen, Research year student, medical student, Aarhus University Hospital
Other Study IDs: 1-10-72-321-12; 2007-58-0010 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2012-07-31; First posted 2012-08-06 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Streptococcal Acute Tonsillitis
Keywords: Acute tonsillitis; Procalcitonin; Streptococcal antigen test; Centor Criteria; Infection marker

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients with acute tonsillitis:
  * Oral temperature, streptococcal rapid antigen detection test, Tonsil surface swab for microbiological culture and a blood sample (measuring the infection markers: Procalcitonin, C-reactive protein, White blood cell count and Absolute neutrophile count).
  Healthy control patients:
  * Tonsil surface swab for microbiological culture.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Acute tonsillitis: Patients with acute tonsillitis aged 15 to 40 years meeting at least two of Centors criteria.
- Healthy control patients: Control patients aged 15 to 40 years.

SUMMARY:
The primary purpose of the present study is to investigate the usefulness of Procalcitonin as a supplement to the Streptococcal antigen test and Centor criteria in the differential diagnose making between Streptococcal and non-Streptococcal acute tonsillitis.

Furthermore, the investigators aim to examine Procalcitonin as a diagnostic marker in acute tonsillitis due to Fusobacterium Necrophorum.

DETAILED DESCRIPTION:
Acute tonsillitis is based on typical symptoms (sore throat, pain on swallowing, and fever) and clinical findings of tonsillar exudate and hyperemia.

10-20% of patients seen by their family physician, have acute tonsillitis due to streptococci group A. In Denmark, Centors criteria and the Streptococcal antigen test (Strep. A-test) are gold standard in the diagnostic process of streptococcal acute tonsillitis. Although the sensitivity and specificity of the Strep. A-test is biochemically high, its clinical reliability is reduced due to several influential factors. Moreover, studies suggest that 4-10% of patients are tested false-negative based on clinical criteria and the Strep A-test.

Fusobacterium necrophorum are suspected to be the cause of acute tonsillitis in teenagers and young adults (5-15%). However, there is no rapid test available for this bacterium. Since tonsillar surface swab is not included in the diagnostic standard, family physicians get no information about infection due to Fusobacterium necrophorum or other pathogens.

C-reactive protein, leukocyte count and absolute neutrophil count as diagnostic markers are examined with variable results. Procalcitonin is a relatively new marker of bacterial infection, which has the advantage of more rapid and specific induction compared to the other markers.

ELIGIBILITY:
Patients with acute tonsillitis:

Inclusion Criteria:

* Age between 15 and 40 years.
* Subjective and objective signs of Acute Tonsillitis + presents of 2-4 Centor Criteria.
* participation accept after verbal and written information.

Exclusion Criteria:

* Antibiotic treatment within the last month.
* Other infection within the last month.
* Inadequate tonsil swabs due to lack of cooperation.
* Suspicion of peritonsillar abscess

Control patients:

Inclusion criteria:

* Age between 15 and 40 years.
* Participation accept after verbal and written information.

Exclusion Criteria:

* Antibiotic treatment within the last month.
* Infection within the last month.
* Tonsillectomy
* More than 2 cases of acute tonsillitis within the last 12 months.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute tonsillitis aged 15 to 40 years consulting their general practitioner with signs and symptoms of acute tonsillitis meeting to or more of Centors criteria.
  Healthy control patients aged 15 to 40 years consulting their general practitioner in other reason than infection.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Procalcitonin | The participants will bee examined in family practice in 30 minuts, measurement results will be available after 3-4 month (average)
  Procalcitonin from all 100 participants will be analyzed at once.

SECONDARY OUTCOMES:
Centor score | The participants will bee examined in family practice in 30 minuts, measurement results will be available after the consultation

OTHER OUTCOMES:
Cultured bacteria | Tonsillar surface swabs obtained at time of consultation. The consultation takes about 30 minuts and results will be analyzed approx. 1 time per week.
  In both the acute tonsillitis group and the healthy control group.

CONTACTS AND LOCATIONS:
Overall Officials: Tejs E Klug, MD, Study Director — Aarhus University Hospital; Therese Ovesen, DMSc, Study Director — Aarhus University Hospital
Locations (1):
- Skoedstrup Medical Clinics, Skødstrup, Denmark

REFERENCES:
- [Result] Elsammak M, Hanna H, Ghazal A, Edeen FB, Kandil M. Diagnostic value of serum procalcitonin and C-reactive protein in Egyptian children with streptococcal tonsillopharyngitis. Pediatr Infect Dis J. 2006 Feb;25(2):174-6. doi: 10.1097/01.inf.0000199273.37314.b2. PMID 16462299
- [Result] Ehlers Klug T, Rusan M, Fuursted K, Ovesen T. Fusobacterium necrophorum: most prevalent pathogen in peritonsillar abscess in Denmark. Clin Infect Dis. 2009 Nov 15;49(10):1467-72. doi: 10.1086/644616. PMID 19842975
- [Result] Diamantis PK, George S, Alexander DK, Georgios MF, Constantinos AB, Sofia M, John AP, George AV. C-Reactive Protein and serum Procalcitonin Levels as Markers of Bacterial Upper Respiratory Tract Infections. American Journal if Infectious Diseases 5(4): 282-287, 2009.
- [Result] Stenfeldt K, Hermansson A. Acute mastoiditis in southern Sweden: a study of occurrence and clinical course of acute mastoiditis before and after introduction of new treatment recommendations for AOM. Eur Arch Otorhinolaryngol. 2010 Dec;267(12):1855-61. doi: 10.1007/s00405-010-1325-9. Epub 2010 Jul 8. PMID 20614127
- [Result] Ylikoski J, Karjalainen J. Acute tonsillitis in young men: etiological agents and their differentiation. Scand J Infect Dis. 1989;21(2):169-74. doi: 10.3109/00365548909039965. PMID 2543062
- [Result] Komaroff AL, Pass TM, Aronson MD, Ervin CT, Cretin S, Winickoff RN, Branch WT Jr. The prediction of streptococcal pharyngitis in adults. J Gen Intern Med. 1986 Jan-Feb;1(1):1-7. doi: 10.1007/BF02596317. PMID 3534166
- [Result] McIsaac WJ, Goel V, To T, Low DE. The validity of a sore throat score in family practice. CMAJ. 2000 Oct 3;163(7):811-5. PMID 11033707
- [Result] Rimoin AW, Walker CL, Hamza HS, Elminawi N, Ghafar HA, Vince A, da Cunha AL, Qazi S, Gardovska D, Steinhoff MC. The utility of rapid antigen detection testing for the diagnosis of streptococcal pharyngitis in low-resource settings. Int J Infect Dis. 2010 Dec;14(12):e1048-53. doi: 10.1016/j.ijid.2010.02.2269. Epub 2010 Oct 30. PMID 21036645
- [Result] Begovac J, Bobinac E, Benic B, Desnica B, Maretic T, Basnec A, Kuzmanovic N. Asymptomatic pharyngeal carriage of beta-haemolytic streptococci and streptococcal pharyngitis among patients at an urban hospital in Croatia. Eur J Epidemiol. 1993 Jul;9(4):405-10. doi: 10.1007/BF00157398. PMID 8243596
- [Result] Lindbaek M, Hoiby EA, Lermark G, Steinsholt IM, Hjortdahl P. Which is the best method to trace group A streptococci in sore throat patients: culture or GAS antigen test? Scand J Prim Health Care. 2004 Dec;22(4):233-8. doi: 10.1080/02813430410006675. PMID 15765639
- [Result] Edmonson MB, Farwell KR. Relationship between the clinical likelihood of group a streptococcal pharyngitis and the sensitivity of a rapid antigen-detection test in a pediatric practice. Pediatrics. 2005 Feb;115(2):280-5. doi: 10.1542/peds.2004-0907. PMID 15687433
- [Result] Del Mar CB, Glasziou PP, Spinks AB. Antibiotics for sore throat. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD000023. doi: 10.1002/14651858.CD000023.pub3. PMID 17054126
- [Result] Rusan M, Klug TE, Ovesen T. An overview of the microbiology of acute ear, nose and throat infections requiring hospitalisation. Eur J Clin Microbiol Infect Dis. 2009 Mar;28(3):243-51. doi: 10.1007/s10096-008-0619-y. Epub 2008 Oct 2. PMID 18830726
- [Result] Aliyu SH, Marriott RK, Curran MD, Parmar S, Bentley N, Brown NM, Brazier JS, Ludlam H. Real-time PCR investigation into the importance of Fusobacterium necrophorum as a cause of acute pharyngitis in general practice. J Med Microbiol. 2004 Oct;53(Pt 10):1029-1035. doi: 10.1099/jmm.0.45648-0. PMID 15358827
- [Result] Jensen A, Hagelskjaer Kristensen L, Prag J. Detection of Fusobacterium necrophorum subsp. funduliforme in tonsillitis in young adults by real-time PCR. Clin Microbiol Infect. 2007 Jul;13(7):695-701. doi: 10.1111/j.1469-0691.2007.01719.x. Epub 2007 Apr 2. PMID 17403128
- [Result] Centor RM. Expand the pharyngitis paradigm for adolescents and young adults. Ann Intern Med. 2009 Dec 1;151(11):812-5. doi: 10.7326/0003-4819-151-11-200912010-00011. PMID 19949147
- [Result] Veasy LG, Tani LY, Hill HR. Persistence of acute rheumatic fever in the intermountain area of the United States. J Pediatr. 1994 Jan;124(1):9-16. doi: 10.1016/s0022-3476(94)70247-0. PMID 7802743
- [Result] Gulich MS, Matschiner A, Gluck R, Zeitler HP. Improving diagnostic accuracy of bacterial pharyngitis by near patient measurement of C-reactive protein (CRP). Br J Gen Pract. 1999 Feb;49(439):119-21. PMID 10326264
- [Result] Kaplan EL, Wannamaker LW. C-reactive protein in streptococcal pharyngitis. Pediatrics. 1977 Jul;60(1):28-32. PMID 327423
- [Result] Putto A, Meurman O, Ruuskanen O. C-reactive protein in the differentiation of adenoviral, Epstein-Barr viral and streptococcal tonsillitis in children. Eur J Pediatr. 1986 Aug;145(3):204-6. doi: 10.1007/BF00446066. PMID 3021463
- [Result] Centor RM, Witherspoon JM, Dalton HP, Brody CE, Link K. The diagnosis of strep throat in adults in the emergency room. Med Decis Making. 1981;1(3):239-46. doi: 10.1177/0272989X8100100304. PMID 6763125
- [Result] Murray PR, Baron EJ, Jorgensen JH, et al. Manual of clinical microbiology. 9th ed. Washington, DC: ASM Press. 2007.